CLINICAL TRIAL: NCT00264446
Title: Phase 1 Study of the Evaluation of Dihydropyrimidine Dehydrogenase (DPD), Uridine Phosphorylase (UP), Orotate Phosphoribosyl Transferase (OPRT), and Thymidine Phosphorylase (TP) Activity in Tissue Resected From Subjects Undergoing Planned Resection of Primary or Metastatic Colorectal Cancer and Liver Biopsy, or Planned Hepatic Resection, Following Administration of Oral ADH300004 (Adherex Protocol Number AHX-03-101)
Brief Title: A Study of ADH300004 in Surgically Resected Primary or Metastatic Colorectal Cancer and Liver Biopsy, or Planned Hepatic Resection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adherex Technologies, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adherex Protocol # AHX-03-101
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2007-08-06 (Estimated); Status verified 2007-08

CONDITIONS: Neoplasms
Keywords: Cancer; Tumors; Neoplasms; Anticarcinogenic Agents; Antineoplastic Agents;; Dihydrouracil dehydrogenase (NADP); Colorectal Carcinoma; Liver Cancer
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Liver Neoplasms | interventions — eniluracil

INTERVENTIONS:
Drug: ADH300004

SUMMARY:
5 fluorouracil (5 FU), one of the most actively investigated anti-cancer drugs, is rapidly inactivated by the enzyme dihydropyrimidine dehydrogenase (DPD). ADH300004 blocks DPD. This study will examine the kinetics of inhibition and recovery of the metabolic pathways for fluoropyrimidines in subjects who receive a single oral dose of ADH300004, and may allow optimization of oral 5 FU dosing to subjects in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* > or = 19 years of age
* Patients with histologically confirmed:

  * primary or metastatic (known or suspected) colorectal carcinoma requiring planned surgical resection with hepatic biopsy and systemic chemotherapy , or
  * primary or metastatic neoplastic disease within the liver from any origin requiring planned surgical resection and systemic chemotherapy
* Adequate performance status and organ function, as evidenced by hematological and biochemical blood testing

Exclusion Criteria:

* Lack of known or suspected metastatic disease in the liver
* Known DPD deficiency
* Severe infection
* Inability to take oral medication
* The need for treatment with any fluoropyrimidine within 8 weeks of any ADH300004 dose
* Stroke, major surgery, or other major tissue injury within 30 days before study entry

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heslin, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB - Division of Surgery, Birmingham, Alabama, United States

REFERENCES:
- See also: Adherex Technologies Inc. Corporate Homepage — http://www.adherex.com